CLINICAL TRIAL: NCT06663384
Title: A Prospective Study Using Augmented Reality Versus Conventional Jig Controls in Total Knee Arthroplasty for Osteoarthritis
Brief Title: ARVIS TKA vs Conventional TKA
Acronym: ARVIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation for Orthopaedic Research and Education (Other)
Collaborators: DonJoy Orthopedics (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: FORE092024
Record Dates: First submitted 2024-10-24; First posted 2024-10-29 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis of knee, Total Knee Replacement
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARVIS arm (Experimental): TKA using ARVIS software
  Interventions: Other: Evaluation of Augmented Reality technology in TKA compared to standard TKA
- conventional TKA (Placebo Comparator): Conventional Total Knee Arthroplasty
  Interventions: Other: Evaluation of Augmented Reality technology in TKA compared to standard TKA

INTERVENTIONS:
Other: Evaluation of Augmented Reality technology in TKA compared to standard TKA — Evaluation of effectiveness of AR system used to perform bone cuts when compared to traditional jigs in primary TKA

SUMMARY:
This study is a pilot analysis of a novel augmented reality guidance platform, the augmented reality visualization and information system (ARVIS, Insight Medical), with aims to demonstrate accuracy of bone resection and implant alignment during kinematic alignment total knee arthroplasty.

DETAILED DESCRIPTION:
This study is a Randomized Controlled Trial evaluating the effectiveness of an AR system utilized to perform bone cuts when compared to traditional jigs in primary TKA for treatment of primary osteoarthritis. Our primary objective is to determine if the ARVIS augmented reality platform is a reliable tool to restore native lower extremity alignment during TKA. An estimated 50 patients will be enrolled in the study, with 25 in the AR-group and 25 in the non-AR conventional kinematic alignment group. A 20% attrition rate (10 patients) is expected throughout the study, leaving 20 patients in each study group. The Investigator intend to evaluate only patients who've met the clinical and radiographic indications for TKA for one knee (Killgren Lawrence Grade > III) and have less than Killgren Lawrence Grade II OA of the contralateral knee. The Investigators intend to use the uninvolved knee as a radiographic comparison to determine ARVIS's post-operative restorative accuracy to the patient's native alignment. Pre- and post-operative radiographs will include standing knee AP, PA, lateral, sunrise, and hip-to-ankle radiographs.

The investigators have chosen to reproduce the patient's native alignment during TKA rather than mechanical alignment given the predominance of recent literature demonstrating superior function and outcome of kinematic based techniques. Intraoperatively, the investigators will use ARVIS to prospectively record bone resection thickness, distal femoral resection angle, femoral component sagittal orientation, femoral component rotation, tibial resection thickness, coronal tibial resection angle, and tibial slope.

The ARVIS is an augmented reality headset with a heads-up display capable of presenting pre-resection hip center and lower extremity alignment. The heads-up display provides real time, intra-operative feedback during bone resections to optimize the component position and lower extremity alignment as compared to the uninvolved contralateral limb. Unlike other methods used to prepare bone cuts during TKA, such as traditional jigs or robotic systems, ARVIS is a self-contained, wearable surgical guidance device controlled by the surgeon, designed to ensure surgeon can focus on their patient while they perform bone cuts on tibia and femur - not a screen across the room.

The procedure of TKA is the same for traditional approach utilizing jigs and ARVIS approach.

ARVIS has received 510(k) clearance from the FDA as of July 2021.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old
* Scheduled for primary conventional TKA with kinematic alignment
* Primary Diagnosis of Osteoarthritis (Killgren Lawrence Grade > III) on affected side
* Able to provide informed consent

Exclusion Criteria:

1. Patients with a previous operation of the same knee, including ACL reconstruction, fracture fixation, previous arthroplasty.
2. Patients that had a conversion to a different procedure intraoperatively or shortly after the TKA.
3. Diagnosed with greater than Killgren Lawrence Grade II OA on the contralateral knee
4. Patients that did not complete the TKA.
5. Patients the Investigator deems not able to follow through with study requirements such as follow-up visits or PROM's.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Radiographic Measurements bilateral knees | From enrollment until 1 year follow-up visit.
  Weight bearing anterposterior (AP), lateral and sunrise views of both knees to measure tibial slope, hip-knee alignment, medial proximal tibial angle, mechanical lateral distal femoral angle, joint line convergence angle, anatomic- mechanical angle.

SECONDARY OUTCOMES:
PROMIS-10 Survey | frome enrollment until 12 month final study visit
  Patient Reported Outcome Measure Information System with 10 questions about subjects pain and function.
Knee Society Score (KSS) | From enrollment until final visit at 12 months after surgery
  A simple and objective scoring system to rate the knee and patient's functional abilities before and after total knee arthroplasty.
Knee Injury and Osteoarthritis outcome Score (KOOS) | from enrollment until completion of study at 12 months post surgery
  KOOS is a 42-item questionnaire that assesses the patient's opinion about the health, symptoms, and functionality of their knee.
Numeric Pain Rating Score (NPRS) | From enrollment until final study visit at 12 months post surgery
  1-10 numeric scale that asks patients to rate their pain in the last 24 hours.

OTHER OUTCOMES:
Virtual Reality Sickness Questionnaire (VSRQ) | After the surgical procedure - one time only
  A motion sickness measurement index specialized in VR environments. 16 questions broken down into three categories (nausea, oculomotor, and disorientation) to assess the severity of each potential cybersickness symptom.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Palumbo, MD, Principal Investigator — Florida Orthopaedic Institute
Locations (1):
- Florida Orthopaedic Institute, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No
This is a pilot analysis of a novel augmented reality guidance platform, the augmented reality visualization and information system (ARVIS, Insight Medical), with aims to demonstrate accuracy of bone resection and implant alignment during kinematic alignment total knee arthroplasty.